CLINICAL TRIAL: NCT05672875
Title: Clinical Specificity Evaluation of the SRI B. Anthracis Lethal Factor Diagnostic System
Brief Title: Evaluation of the SRI B. Anthracis Lethal Factor Diagnostic System
Status: Terminated | Type: Observational
Why Stopped: Sponsor decision
Sponsor: SRI International (Industry)
Collaborators: Department of Health and Human Services (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: 4650.367
Record Dates: First submitted 2023-01-03; First posted 2023-01-05 (Actual); Last update posted 2023-11-30 (Actual); Status verified 2023-11

CONDITIONS: Anthrax
MeSH Terms: conditions — Anthrax

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Healthy and Symptomatic Subjects: Blood sample testing on the Anthrax LF Dx System
  Interventions: Diagnostic Test: Anthrax LF Dx System

INTERVENTIONS:
Diagnostic Test: Anthrax LF Dx System — Lateral flow immunoassay for the detection of the LF biomarker in whole blood samples.

SUMMARY:
This study is intended to estimate the Anthrax LF Dx System specificity. Sensitivity will be estimated with 10% of the samples spiked with recombinant Bacillus anthracis lethal factor (LF) used to prepare contrived positive samples.

DETAILED DESCRIPTION:
This is a prospective, non-interventional, multi-center study assessing the clinical specificity of the Anthrax LF Dx System using venous blood samples collected from presumptive anthrax negative adult male and female healthy and symptomatic subjects (non- B. anthracis infected).

Up to 500 subjects may be enrolled to meet the goal of 440 evaluable subjects (220 healthy and 220 symptomatic). Subjects will have one venous blood sample collected from a single time-point tested with the Anthrax LF Dx System. At each clinical site, specimens will be randomly selected such that 10% (40 of 400) of all subjects' venous blood samples (total of 40 [20 healthy and 20 symptomatic]) will be spiked with recombinant B. anthracis LF to prepare a contrived positive sample. An unblinded operator will prepare the spiked samples and provide both the spiked and neat samples to a blinded operator for testing on the Anthrax LF Dx System. Thus, the blinded operator will receive samples that could either be spiked (positive) or neat (presumed negative) to preserve the blind.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subject who is ≥18 years of age
* Subject is willing and able to provide Informed Consent for study participation, prior to any study mandated procedures
* For the healthy human population: Subject is in general good health with a stable health status based on medical history, and the investigator's clinical judgment defined as:

  * No acute medical conditions that require the use of systemic prescription medications in the last 30 days and
  * Any chronic medical diagnoses/conditions should be stable for the last 30 days (no hospitalizations, emergency room (ER), or urgent care for condition). This includes no change in chronic prescription medication, dose, or frequency as a result of deterioration of the chronic medical diagnosis/condition in the 30 days before enrollment.
* For the symptomatic human population:

  * Current symptoms consistent with cold, flu or other bronchial and symptomatic infections. The subject must currently (day of consent) have at least one of the following symptoms: fever, chills, chest discomfort, shortness of breath, cough, dizziness/confusion, nausea, headache, sweats, fatigue, or body aches.

Exclusion Criteria:

* Subject has inclusion symptoms and tests positive for COVID-19.
* Subject has previously enrolled in this study, or subject has previously failed screening for this study.
* Subject has any medical or social or psychiatric condition(s) or current substance abuse that, in the opinion of the investigator, would preclude the subject's ability to provide informed consent/assent, or to comply with the study requirements.
* Currently enrolled in an investigational drug or device clinical study in which the primary endpoint has not occurred or occurred within the last 30 days.
* Subject is a nursing home resident.
* Subject is a prisoner.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult male and female healthy and symptomatic subjects.
Sampling Method: Probability Sample
Enrollment: 343 (Actual)
Dates: Start 2023-01-23 (Actual); Primary Completion 2023-04-20 (Actual); Study Completion 2023-04-20 (Actual)

PRIMARY OUTCOMES:
The estimated negative percent agreement (NPA) of the Anthrax LF Dx System test. | Day of enrollment
  The estimated NPA will be calculated from testing neat specimens from 400 subjects (with presumed negative samples).
Adverse events | Within 24 hours of blood draw
  All adverse events directly related to specimen collection will be reported.

SECONDARY OUTCOMES:
The estimated percent positive agreement (PPA) of the Anthrax LF Dx System test. | Day of enrollment
  PPA will be estimated with samples spiked with recombinant B. anthracis lethal factor (LF) used to prepare contrived positive samples.

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - WellNow Urgent Care and Research, Cincinnati, Ohio
  - WellNow Urgent Care and Research, Columbus, Ohio
  - WellNow Urgent Care and Research, Dayton, Ohio

IPD SHARING:
Plan to Share IPD: Undecided